CLINICAL TRIAL: NCT00605345
Title: An Open Label Randomised Controlled Study to Compare the Efficacy, Safety and Tolerability of Once-monthly Administration of Subcutaneous Mircera Versus Darboepoetin Alfa for the Maintenance of Haemoglobin Levels in Renal Transplant Recipients With Chronic Renal Anaemia.
Brief Title: A Study Comparing Subcutaneous Mircera and Darbepoetin Alfa for Maintenance Treatment of Anemia in Kidney Transplant Recipients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML21058
Record Dates: First submitted 2008-01-18; First posted 2008-01-31 (Estimated); Results first posted 2016-08-05 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-04

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — Darbepoetin alfa; continuous erythropoietin receptor activator

ARMS (2):
- CERA Treatment Once Monthly (Experimental)
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]
- Darbepoetin Alfa Once Biweekly (Active Comparator)
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: Darbepoetin alfa — As prescribed
  Arms: Darbepoetin Alfa Once Biweekly
Drug: methoxy polyethylene glycol-epoetin beta [Mircera] — 120, 200 or 360 micrograms sc 4-weekly (starting dose)
  Arms: CERA Treatment Once Monthly

SUMMARY:
This two arm study will compare the efficacy and safety of subcutaneous Mircera versus darbepoetin alfa for the maintenance of hemoglobin levels in kidney transplant recipients with chronic renal anemia. Patients currently receiving maintenance treatment with darbepoetin alfa will be randomized either to receive 4-weekly injections of Mircera with a starting dose (120, 200 or 360 micrograms subcutaneously) derived from the dose of darbepoetin alfa they were receiving in the 2 weeks preceding study start, or to stay on 2-weekly darbepoetin alfa therapy. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, > or = 18 years of age;
* kidney transplant recipients with stage 3 or stage 4 chronic kidney disease;
* functioning graft of > 6 months and < 10 years after kidney transplantation, with no signs of acute rejection;
* stable maintenance subcutaneous darbepoetin alfa therapy every 2 weeks.

Exclusion Criteria:

* transfusion of red blood cells during previous 2 months;
* poorly controlled hypertension;
* significant acute or chronic bleeding;
* need for dialysis therapy expected in next 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2007-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (16):
- Spain (16):
  - Alicante, Alicante
  - Badajoz, Badajoz
  - Badalona, Barcelona
  - Barcelona, Barcelona
  - L'Hospitalet de Llobregat, Barcelona
  - Santander, Cantabria
  - Ciudad Real, Ciudad Real
  - Córdoba, Cordoba
  - Granada, Granada
  - A Coruña, La Coruña
  - Santiago de Compostela, La Coruña
  - Madrid, Madrid
  - Valencia, Valencia
  - Valladolid, Valladolid
  - Barakaldo, Vizcaya
  - Galdakao, Vizcaya

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280
- [Derived] Campistol JM, Carreno A, Morales JM, Pallardo L, Franco A, Navarro D, Grinyo JM, Montenegro J, Sanchez Fructuoso AI, Romero R, Guirado L, Arias M; TIVOLI Study Group. Once-monthly pegylated epoetin Beta versus darbepoetin alfa every two weeks in renal transplant recipients: a randomized trial. Transplantation. 2013 Jan 27;95(2):e6-e10. doi: 10.1097/TP.0b013e3182782f3a. No abstract available. PMID 23325012

RESULTS

PARTICIPANT FLOW:
Groups:
- CERA Treatment Once Monthly: CERA 120, 200 or 360 micrograms subcutaneously
- Darbepoetin Alfa Once Biweekly: Darbepoetin Alfa as prescribed
Period: Overall Study
Arm/Group | CERA Treatment Once Monthly | Darbepoetin Alfa Once Biweekly
Started | 46 | 25
Completed | 45 | 22
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CERA Treatment Once Monthly | Darbepoetin Alfa Once Biweekly | Total
Number analyzed (Participants) | 46 | 25 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (11.04) | 56.7 (10.49) | 55.3 (10.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 8 | 35
  Male | 19 | 17 | 36
Region of Enrollment [Number; unit: participants]
  Spain | 46 | 25 | 71

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants Maintaining Average Haemoglobin (Hb) Concentration During the Efficacy Evaluation Period (EEP) Within the Target Range
Description: Key outcomes will be assessed during the first 12 weeks following the 16 weeks dose titration period, i.e. during the Efficacy Evaluation Period (EEP). Assessments performed every four weeks, beginning at week 16 up to week 28. The reference haemoglobin is defined as the mean of the two assessments recorded during the SVP (weeks -4 and -2). For the purposes of efficacy assessment the target haemoglobin concentration range will be defined as ± 1 g/dL of the reference haemoglobin concentration AND within the range 10 - 12 g/dL.
Time Frame: Weeks 16-28
Population: Analysis was performed in the per protocol (PP) population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CERA Treatment Once Monthly | Darbepoetin Alfa Once Biweekly
Number analyzed (Participants) | 42 | 21
percentage of participants | 64.29 [48.03 to 78.45] | 57.14 [34.02 to 78.18]
Statistical Analysis 1: Comparison: CERA Treatment Once Monthly vs Darbepoetin Alfa Once Biweekly; Test type: Non-Inferiority or Equivalence — Non-inferiority was met if the lower limit of the confidence interval for the response rate of the CERA group was greater than the observed response rate of the darbepoetin group minus 15%. The calculated lower limit of an acceptable difference in response rates thus, was based on the actual percentage of "responders" in the darbepoetin group and this percentage minus 15% had to be excluded; p = 0.5947, Fisher Exact

2. Secondary Outcome: Mean Change in Hb Concentration From Baseline to Efficacy Evaluation Period (EEP)
Description: Reference haemoglobin at baseline is defined as the mean of the two assessments recorded at weeks -4 and -2. Additional assessments were then performed every 4 weeks at week 0 through week 28. Mean change was calculated as value at 28 weeks minus baseline.
Time Frame: Baseline to 28 weeks
Population: Analysis performed in the Intent toTreat (ITT) population, which includes all participants receiving at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | CERA Treatment Once Monthly | Darbepoetin Alfa Once Biweekly
Number analyzed (Participants) | 46 | 25
g/dL | 0.08 (0.85) | 0.05 (1.06)

3. Secondary Outcome: Percentage of Participants Maintaining Hb Concentration in 10-12 g/dL Range Throughout the Efficacy Evaluation Period (EEP)
Time Frame: Weeks 16-28
Population: Analysis performed with intent to treat (ITT) population, which includes all participants receiving at least one dose of the study drug.
Measure: Number; unit: percentage of participants
Arm/Group | CERA Treatment Once Monthly | Darbepoetin Alfa Once Biweekly
Number analyzed (Participants) | 46 | 25
percentage of participants | 71.7 | 64.0

4. Secondary Outcome: Mean Time Spent in 10-12g/dL Range During the Efficacy Evaluation Period (EEP)
Description: Efficacy Evaluation Period was the 12 weeks following 16 weeks of treatment in the Dose Titration Period.
Time Frame: Weeks 16-28
Population: Analysis was performed using the intent to treat (ITT) population, which includes all participants receiving at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CERA Treatment Once Monthly | Darbepoetin Alfa Once Biweekly
Number analyzed (Participants) | 46 | 25
days | 57.0 (23.98) | 50.5 (27.7)

5. Secondary Outcome: Percentage of Participants Needing Dose Adjustments
Description: Assessment of the Dose Titration Period of 16 weeks of treatment and following 12 weeks, known as the Efficacy Evaluation Period (EEP).
Time Frame: Up to 28 weeks
Population: Analysis was performed on the safety population.
Measure: Number; unit: percentage of participants
Arm/Group | CERA Treatment Once Monthly | Darbepoetin Alfa Once Biweekly
Number analyzed (Participants) | 46 | 25
percentage of participants
  Dose Titration Period | 73.9 | 56.0
  Efficacy Evaluation Period (n=45,23) | 33.3 | 20.8

6. Secondary Outcome: Incidence of RBC Transfusions
Description: as for outcome 5
Time Frame: Up to 28 weeks
Population: Analysis performed with the intent to treat (ITT) population, which includes all participants receiving at least one dose of the study drug.
Measure: Number; unit: participants
Arm/Group | CERA Treatment Once Monthly | Darbepoetin Alfa Once Biweekly
Number analyzed (Participants) | 46 | 25
participants | 1 | 2

ADVERSE EVENTS:
Time Frame: Up to 28 weeks
Description: The intent to treat (ITT) population included all participants receiving at least one dose of the study drug. This population was primarily used for the reporting of safety information.
Arm/Group | CERA Treatment Once Monthly | Darbepoetin Alfa Once Biweekly
Serious Adverse Events (participants affected / at risk) | 9/46 | 3/25
Other Adverse Events (participants affected / at risk) | 27/46 | 16/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CERA Treatment Once Monthly (N=46) | Darbepoetin Alfa Once Biweekly (N=25)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 2 (3) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Device Breakage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Laryngeal Granuloma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aneurysm (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CERA Treatment Once Monthly (N=46) | Darbepoetin Alfa Once Biweekly (N=25)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 2 (2)
Asthenia (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 3 (3)
Oedema (General disorders) | 2 (2) | 2 (2)
Oedema Peripheral (General disorders) | 3 (3) | 3 (3)
Escherichia Urinary Tract Infection (Infections and infestations) | 5 (5) | 0 (0)
Influenza (Infections and infestations) | 3 (4) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 4 (4)
Upper Respiratory Tract Infection (Infections and infestations) | 6 (6) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 4 (4) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 9 (9) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.